CLINICAL TRIAL: NCT06750653
Title: Skin Barrier Function and Inflammation in Aging: The BIA Study
Acronym: BIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-34535; R21AR082620 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Inflammation; Skin Inflammation; Aging
Keywords: CeraVe; Vaseline; Aging; Inflammation; Skin; Older Adults
MeSH Terms: conditions — Inflammation; Dermatitis | interventions — Petrolatum

STUDY DESIGN:
Intervention Model Description: Subjects will act as their own control - they will be asked to apply the study moisturizer they are randomized to for one intervention period (4 weeks) and not to apply topical moisturizers for the other 4- week intervention period).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Access to the randomization code will be strictly controlled.
  The moisturizing products will be placed in identical cardboard boxes by a staff member not involved in the disease assessments so that investigators taking assessments will not be aware of which study arm participants were randomized to. Participants will be asked not to open the cardboard packaging until they leave the study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CeraVe First (Active Comparator): CeraVe for 4 weeks; then no moisturizer for 4 weeks. CeraVe Moisturizing Cream containing ceramides and hyaluronic acid manufactured by L'Oréal, for topical skin use.
  Interventions: Other: CeraVe Moisturizing Cream
- CeraVe Second (Active Comparator): No moisturizer for 4 weeks, then CeraVe for the second 4-week study period. CeraVe Moisturizing Cream containing ceramides and hyaluronic acid manufactured by L'Oréal, for topical skin use
  Interventions: Other: CeraVe Moisturizing Cream
- Vaseline First (Active Comparator): Vaseline for 4 weeks then no moisturizer for 4 weeks. Vaseline white petrolatum, manufactured by Unilever, for topical skin use.
  Interventions: Drug: Vaseline
- Vaseline Second (Active Comparator): No moisturizer for 4 weeks; then Vaseline for 4 weeks. Vaseline white petrolatum, manufactured by Unilever, for topical skin use.
  Interventions: Drug: Vaseline

INTERVENTIONS:
Other: CeraVe Moisturizing Cream — CeraVe is a formulation of Purified Water, Glycerin, Cetareth-20 and Cetearyl Alcohol, Caprylic/Capric Triglyceride, Behentrimonium Methosulfate and Cetearyl Alcohol, Cetyl Alcohol, Petrolatum, Dimethicone, Hyaluronic Acid, Ceramide 1, Ceramide 3, Ceramide 6-II, Cholesterol, Phytosphingosine, Potassium Phosphate, Dipotassium phosphate, Phenoxyethanol, Methylparaben, Propylparaben, Disodium EDTA, Sodium Lauroyl Lactylate, Carbomer, Xanthan Gum, manufactured by L'Oréal, for topical skin use.
  Arms: CeraVe First; CeraVe Second
Drug: Vaseline — Vaseline is a formulation of active ingredient white petrolatum, USP (100%), manufactured by Unilever, for topical skin use.
  Arms: Vaseline First; Vaseline Second

SUMMARY:
This is a randomized, investigator-blinded, self-controlled pilot study of the physiologic response to topical moisturizers among older adults with dry skin. The overarching hypothesis is that skin barrier decline is an important source of chronic inflammation, and that skin barrier restoration with moisturizers can reduce serum biomarkers of inflammation. The primary objective is to determine the feasibility for a larger trial, and the secondary objectives are to determine the extent to which measures of serum inflammation, skin barrier function, and the skin microbiome change in response to moisturizers. Participants will be asked to apply one of two topical moisturizers that are widely available over the counter in the US (Vaseline® 100% pure petroleum jelly or CeraVe® moisturizing cream) once daily for 4 weeks to the front of the torso, buttocks, arms, and legs. Subjects will act as their own control (i.e. they will be asked to apply the study moisturizer they are randomized to for one intervention period (4 weeks) and not to apply topical moisturizers for the other 4- week intervention period). Participants will be randomized in a 1:1:1:1 ratio to one of 4 treatment groups: i. no intervention then CeraVe; ii. CeraVe then no intervention; iii. no intervention then Vaseline; iv. Vaseline then no intervention. At each visit (baseline, week 4, and week 8), participants will undergo skin barrier testing, skin microbiome sampling, and phlebotomy to measure serum inflammatory markers.

DETAILED DESCRIPTION:
In older adults, inflammation is associated with geriatric conditions, including multimorbidity and frailty, that result in premature death. This phenomenon has been termed 'inflammaging,' and multiple potential mechanisms have been identified, including chronic infections, visceral obesity, increased gut permeability, and cellular senescence, among others.1,2 Limited data suggest that age-associated barrier decline in the skin may also play an important role. Beginning at about age 50, skin barrier decline is caused by decreased Na+/H+ antiporter activity and impaired stratum corneum acidification.3 Persons >70 years of age also suffer from additional defects in cutaneous lipid production.4 The result is reduced resilience to minor injury and epidermal cytokine generation, which may have significant systemic effects, given that the skin is the body's largest organ.5 Additionally, changes in the skin barrier may result in dysbiosis and increased exposure to microbial products, as has been seen in age-associated gut barrier decline.6 Skin barrier decline has been directly correlated with levels of keratinocyte-derived inflammatory markers in aged mice.7 Furthermore, there is experimental evidence that application of moisturizers to aged skin may improve skin barrier function and reduce inflammation. In aged mice, application of petrolatum twice daily for 10 days significantly reduced cutaneous and serum inflammatory cytokines including TNFalpha, IL-1alpha, IL-1beta, and IL-6 after minor injury.7 The investigators propose a randomized, investigator-blinded, self-controlled pilot study of the physiologic response to topical moisturizers among older adults with dry skin. The overarching hypothesis is that skin barrier restoration with moisturizers can reduce serum biomarkers of inflammation. The primary objective is to determine the feasibility for a larger trial, and the secondary objectives are to determine the extent to which measures of serum inflammation, skin barrier function, and the skin microbiome change in response to moisturizers. Participants will be asked to apply one of two topical moisturizers that are widely available over the counter in the US (Vaseline® 100% pure petroleum jelly or CeraVe® moisturizing cream) once daily for 4 weeks to the front of the torso, buttocks, arms, and legs. Subjects will act as their own control (i.e. they will be asked to apply the study moisturizer they are randomized to for one intervention period (4 weeks) and not to apply topical moisturizers for the other 4- week intervention period). Participants will be randomized in a 1:1:1:1 ratio to one of 4 treatment groups: placebo i. no intervention then CeraVe; ii. CeraVe then no intervention; iii. no intervention then Vaseline; iv. Vaseline then no intervention. At each visit (baseline, week 4, and week 8), participants will undergo skin barrier testing, skin microbiome sampling, and phlebotomy to measure serum inflammatory markers.

ELIGIBILITY:
Inclusion Criteria

1. Male or female ≥ 70 years of age at the baseline visit.
2. Diagnosis of xerosis cutis based on an Overall Dry skin (ODS) score of => 1 for any body site where patients will be asked to apply moisturizer (i.e. arms, legs, buttocks, front of trunk).
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative
4. Ability for subject to comply with the requirements of the study.

Exclusion Criteria

1. History of inflammatory skin disease (e.g. psoriasis, atopic dermatitis, or bullous pemphigoid) that has been active in the past 10 years.
2. History of contact dermatitis to moisturizers.
3. History of chronic inflammatory conditions (such as cancer, arthritis, inflammatory bowel disease, or coronary artery disease). Participants with a history of localized skin cancer will not be excluded.
4. Current infection.
5. Open skin wounds.
6. Physical limitations or lack of a caregiver preventing application of a moisturizer to skin on the trunk and extremities.
7. Current use of topical medications, oral systemic immunomodulatory treatments, or anti-microbial treatments.
8. Diagnosis of primary or acquired immunodeficiency.
9. Use of skin moisturizer less than 1 week prior to enrollment visit, with the exception that participants may use non-study moisturizer/sunscreen on face, if used consistently throughout study period.
10. Inability to give informed consent.
11. Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.
12. If the participant does not meet all the above criteria, he/she will not be eligible for study participation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate feasibility | 8 weeks
  To demonstrate the feasibility of a moisturizer-based skin barrier enhancement randomized controlled trial using these measures:
  Enrollment Rate: Number of participants enrolled in the study within a specified time frame
  Retention Rate: Percentage of participants who complete the study without dropping out, assessed at the end of the trial.
  Adherence to Protocol: Percentage of participants who adhere to the treatment regimen as outlined, calculated based on participant self-reports or product usage logs.
  Data Collection Completeness: Percentage of complete data sets collected for the primary outcome measure at baseline and follow-up.

SECONDARY OUTCOMES:
Change in composite inflammation score | 4 weeks
  Mean of the individual z-scores for serum inflammatory markers. Mean of the Individual Z-Scores for Serum Inflammatory Markers" assesses the standardized values (z-scores) of serum inflammatory markers in a population.
  The normal range for z-scores is typically considered to be between:
  -2 and +2: This range typically encompasses about 95% of the data in a normally distributed population.
  Outcome Interpretation: Higher z-scores indicate worse outcomes, as they suggest higher levels of inflammatory markers, which are typically associated with inflammation and various health issues.
Change in skin barrier function | 4 weeks
  Transepidermal water loss.
Change in skin barrier function | 4 weeks
  Changes in skin hydration will be measured and recorded using a Tewameter which quantifies the amount of water that evaporates from the skin's surface. Low TEWL values suggest better skin hydration.
Change in skin barrier function | 4 weeks
  pH.
Change in skin barrier function | 4 weeks
  Skin Electrical Impedance Spectroscopy Device: A specialized device designed for skin analysis that delivers a small-range alternating current to the skin surface and measures the voltage response to determine impedance.
  Low Impedance Values: Generally indicate better skin hydration, as water facilitates increased conductivity.
  High Impedance Values: Suggest lower hydration levels or impaired skin barrier function, as drier skin has reduced conductivity.
Measures of skin microbial composition diversity | 4 weeks
  Differences in overall microbiome composition after moisturizer application

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Abuabara, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide individual participant level data (IPD) in a de-identified format, along with a data dictionary, statistical analysis plan, analytic code, and the final protocol. This data will be available through the Vivli platform, a non-profit organization dedicated to clinical research data sharing. Data access will be granted as soon as possible or at the time of publication and will be preserved for a minimum of five years post-funding.
  All shared data will be de-identified using the safe harbor method, following HIPAA privacy regulations. To access the IPD, users must complete the Vivli data request form and sign the Data Use Agreement, which restricts data use and requires data security. Users must submit a valid scientific question and a statistical analysis plan. Approved requests will receive access to the data at no cost for a designated period, with Vivli ensuring storage and access for as long as the data holds scientific value.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available as soon as possible or at the time of associated publication. The duration of preservation and sharing of the data will be a minimum of 5 years after the end of the funding period.
  The investigators anticipate the IPD will be made available Starting October 1, 2026 through September 30, 2031.
Access Criteria: The investigators will share individual participant level or IPD data. The data will be made available in a de-identified format. The investigators will also share the data dictionary, statistical analysis plan, analytic code, and final protocol with amendments.
  In order to maintain appropriate managed access of the data, the investigators will make it available via the Vivli platform. Vivli is a non-profit clinical research data sharing platform that has been created to meet the needs of researchers who use and produce clinical research data worldwide.
  Anyone who has submitted an approved data request and signed a data use agreement on Vivli will be given access to the data. In order to get access to the data, the user must submit a valid scientific question, include a statistical analysis plan, and complete all required fields on the Vivli data request form.
URL: https://abuabara.ucsf.edu/